CLINICAL TRIAL: NCT05187273
Title: Intraoperative Fluid Optimization Based on a Dynamic Elastance Protocol During Major Abdominal Surgery: a Randomised Control Trial
Brief Title: Hemodynamic Optimization Based on a Dynamic Elastance Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RUSSO ANDREA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: ID3724
Record Dates: First submitted 2021-12-25; First posted 2022-01-11 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Fluid Management

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental)
  Interventions: Behavioral: Elastance Group
- control (No Intervention)

INTERVENTIONS:
Behavioral: Elastance Group — Fluids are given based on dynamic elastane value
  Arms: intervention

SUMMARY:
In this study investigators explore the effects of a dynamic elastance guided protocol compared to a stroke volume variation fluid therapy on lactate levels during major abdominal surgery. Hence investigators created two groups: in the intervention group fluids are given in fluid-responders (SVV > 13%) based on high value of dynamic elastance (ie. Eadyn > 0.9). In the standard group fluids are administered when SVV > 13%.

ELIGIBILITY:
Inclusion Criteria: patients enrolled for major abdominal surgery

-

Exclusion Criteria:

1. end-stage renal disease
2. severe heart dysfunction
3. heart rhythm alterations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
lactate levels | at the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: andrea russo, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli
Locations (1):
- Andrea Russo, Rome, Italy

REFERENCES:
- [Derived] Russo A, Aceto P, Cascarano L, Menga LS, Romano B, Carelli S, Console E, Pugliese F, Cambise C, Fiorillo C, Alfieri S, Antonelli M, Sollazzi L, Dell'Anna AM. A dynamic elastance-based protocol to guide intra-operative fluid management in major abdominal surgery: A randomised clinical trial. Eur J Anaesthesiol. 2025 Aug 1;42(8):727-736. doi: 10.1097/EJA.0000000000002162. Epub 2025 Mar 11. PMID 40070308